CLINICAL TRIAL: NCT00712543
Title: A Preference Study Comparing Kristalose® and Liquid Lactulose in the Treatment of Constipation
Brief Title: A Preference Study Comparing Kristalose® and Liquid Lactulose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KR-001
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-08

CONDITIONS: Constipation
Keywords: constipation; laxative; lactulose; Kristalose®
MeSH Terms: conditions — Constipation | interventions — Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Kristalose®, as prescribed, for 7 days.
  Interventions: Drug: lactulose (Kristalose®)
- 2 (Experimental): Liquid lactulose, as prescribed, for 7 days.
  Interventions: Drug: liquid lactulose

INTERVENTIONS:
Drug: lactulose (Kristalose®) — Crystals to be dissolved in water and taken as prescribed.
  Other Names: Kristalose®
  Arms: 1
Drug: liquid lactulose — Liquid to be taken as prescribed.
  Arms: 2

SUMMARY:
This study will evaluate whether patients have an overall preference for Kristalose® or liquid lactulose based on taste, consistency, and portability.

DETAILED DESCRIPTION:
This study will evaluate whether patients have an overall preference for Kristalose® or liquid lactulose based on taste, consistency, and portability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recently diagnosed chronic constipation requiring treatment.

Exclusion Criteria:

* Patients with galactosemia (galactose-sensitive diet).
* Patients less than 18 years of age.
* Patients currently on lactulose therapy.
* Inability to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]) and agree to abide by the study restrictions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Arya Gastroenterology Associates, Brooklyn, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Rapid Medical Research, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from the outpaient clinics of Wake Research Associates (Raleigh, NC); Rapid Medical Research (Cleveland, OH) and Arya Gastroenterology (Brooklyn, NY) between June 2009 and August 2009.
Groups:
- Powder, Then Liquid Lactulose: Kristalose (powder lactulose), as perscribed, for the first 7 days, then liquid lactulose (as perscribed) for the second 7 days.
- Liquid, Then Powder Lactulose: Liquid lactulose, as perscribed, for the first 7 days, then Kristalose (powder lactulose), as perscribed, for the second 7 days.
Period: Day 1-7
Arm/Group | Powder, Then Liquid Lactulose | Liquid, Then Powder Lactulose
Started | 23 | 27
Completed | 23 | 27
Not Completed | 0 | 0
Period: Day 8-14
Arm/Group | Powder, Then Liquid Lactulose | Liquid, Then Powder Lactulose
Started | 23 | 27
Completed | 23 | 25
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Powder, Then Liquid Lactulose | Liquid, Then Powder Lactulose | Total
Number analyzed (Participants) | 23 | 27 | 50
Age, Customized [Mean (Standard Deviation); unit: years] | 44.02 (13.37) | 52.37 (15.71) | 48.61 (14.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 5 | 8 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 11 | 26
  White | 3 | 10 | 13
  Hispanic | 4 | 5 | 9
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Preference in Terms of Overall Preference and Preference of Taste, Consistency, and Portability.
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Powder, Then Liquid Lactulose | Liquid, Then Powder Lactulose
Number analyzed (Participants) | 23 | 27
participants
  Preferred liquid lactulose overall | 7 | 6
  Preferred powder lactulose overall | 12 | 11
  No preference overall | 4 | 8
  Preferred liquid lactulose in terms of taste | 7 | 9
  Preferred powder lactulose in terms of taste | 12 | 11
  No preference in terms of taste | 4 | 5
  Preferred liquid lactulose in terms of consistency | 7 | 7
  Preferred powder lactulose in terms of consistency | 11 | 11
  No preference in terms of consistency | 5 | 7
  Preferred liquid lactulose in terms of portability | 1 | 4
  Preferred powder lactulose in terms of portability | 17 | 16
  No preference in terms of portability | 5 | 5

ADVERSE EVENTS:
Arm/Group | Powder, Then Liquid Lactulose | Liquid, Then Powder Lactulose
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 13/50 | 10/50
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Powder, Then Liquid Lactulose (N=50) | Liquid, Then Powder Lactulose (N=50)
Flatulence (Gastrointestinal disorders) | 7 (7) | 6 (6)
Abdominal distention (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain, upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain, lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pharyngoleryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Menstrual cramps (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No